CLINICAL TRIAL: NCT03678974
Title: Targeted Healthcare Efforts to Bridge Resources, Improve the Development of Guideline-based Exercise Prescription and Reduce Obesity by Joining Education, Community, and Technology. (THE BRIDGE PROJECT - Pilot Study)
Brief Title: Bridging Resources Improve the Development of Guideline-based Exercise
Acronym: BRIDGE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: Brentwood Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-906
Record Dates: First submitted 2018-08-27; First posted 2018-09-20 (Actual); Last update posted 2020-02-13 (Actual); Status verified 2020-02

CONDITIONS: Obesity; Physical Activity
Keywords: Cardiorespiratory Fitness; Intensive Behavioral Therapy for Obesity; Exercise Prescription
MeSH Terms: conditions — Obesity; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise (Experimental): Subjects will receive metabolic testing, exercise prescription, YMCA memberships, and physician based on Intensive Behavioral Therapy for Obesity utilizing CardioCoach app.
  Interventions: Behavioral: Exercise Prescription

INTERVENTIONS:
Behavioral: Exercise Prescription — The CardioCoach Vo2Max app allows the physician to upload an individual's Vo2 Max and resting metabolic rate results to the app which will allow each subject to view those results in the context of workout zones, goals, and energy balance. The app shows time spent aerobic versus anaerobic, and the actual number of calories burned during a workout and post-workout. It will also show what fuel source (Fats vs Carbs) are being used in real time during your workouts. Subjects can be guided through their workouts utilizing voice coaching to keep you in your customized zones. Additionally, the app accommodates a quick add of calories directly to the app to track calories consumed vs calories burned.

SUMMARY:
The purpose of this pilot study is to more effectively deliver the current standard of care for obesity and physical activity based on current guidelines. The investigators plan to gather preliminary data on physician-directed Intensive Behavioral Therapy for Obesity (IBT-O) utilizing CardioCoachCO2 by KORR technology to measure oxygen consumption both at rest and during exercise to assess resting metabolic rate (RMR) and cardiorespiratory fitness (CRF) respectively. RMR and CRF will be incorporated into an exercise prescription through implementation of the CardioCoach VO2 Max App as part of a multi-level physical activity intervention to improve CRF and decrease obesity by acting on multiple levels of the socio-ecological model in a primary care setting.

DETAILED DESCRIPTION:
Experimental, One-Group Pretest-Posttest study, in which current physical activity levels and cardiorespiratory fitness (CRF) will be evaluated and assessed at baseline and following 6 months of exercise conditioning. Over the course of 6 months (26 weeks) subjects will have physician based follow up appointments based on IBT-O by CMS criteria with the primary outcome of improving CRF by 1 MET, which has been associated with a 12% decrease in mortality. Secondary outcomes will include meeting changes in BMI consistent with CMS criteria of achieving a weight loss of at least 6.6 lbs (3kg) during the first six months of IBT in order to continue with IBT coverage. Progressing patients safely and efficiently toward achieving current physical activity recommendations within a sample population to guide future research on a larger scale. Through questionnaires the investigators will also gather data on Stages of Change Readiness, osteoarthritis of the knee and other weight-bearing joints, and overall Quality of Life. Subjects will be approved by their primary care physician prior to study participation. Based on American College of Sports Medicine (ACSM's) 2015 preparticipation health screening guidelines, if medical clearance is required then subjects will need to make an appointment with their PCP for exercise clearance prior to subjects' first week of participation and prior to any exercise testing. Information collected will included demographic (age, gender, race, occupation, current employment status) and co-morbid medical conditions such as hypertension, diabetes, coronary artery disease, renal disease, heart failure, etc. or any other significant illness.

On the first day of testing subjects after an overnight fast of at least 12 hours for determination of RMR through indirect calorimetry. After completing the RMR assessment, subjects will complete the following instruments: assessment of current physical activity level, Stage of Readiness to Change, personal health goals, screened by symptom assessment and physical examination for osteoarthritis of the knee and other weight-bearing joints, screening for depression and overall Quality of Life through the application of a questionnaires in a primary care setting.

On the 2nd day subjects will perform a symptom limited cardiopulmonary exercise (CPX) testing on a treadmill using a modified Balke protocol. Subjects will each be provided with their own personal heart rate monitor. The initial graded exercise test will be performed with the heart rate monitor being worn. Subjects will keep their own heart rate monitor during the study, and they will wear them during their workouts so that the app can keep them in their target heart rate zone. They will also wear the monitors during their 6 month graded exercise test. After completion of the CPX, Subjects will be instructed on how to download and utilize the CardioCoach VO2 Max app available on Smartphones which is compatible with Polar H10 Heart rate monitor system.

Subjects will be provided with access to the YMCA within their community to implement their exercise prescription.

This IBT-O model utilizing CardioCoachCO2 technology to improve physical activity, will follow the requirements developed by CMS for coverage of an IBT for Obesity

1. One face-to-face visit every week for the first month,
2. One face-to-face visit every other week for months 2-6,
3. At the six-month visit, a reassessment of Obesity and CRF through CPX. A healthy meal plan has been included as part of standard of care based on CMS IBT guidelines. Subjects will be counseled on the development of a healthy meal plan. This healthy meal plan will incorporate each subject's RMR as the foundation for caloric requirements. In addition to being counseled on the development of a healthy meal plan, subjects will be educated and counseled on Intermittent Fasting (IF).

During the study, the investigators will monitor fitness indicators (physical activity level, weight, BMI, BP, resting HR, VO2Peak, VO2Max, RER, Test time, METpeak, HRmax, HRrecovery, calories burned) and adherence (number of sessions performed at YMCA/month compared goal of 12 exercise sessions/4 weeks), in addition to physical activity performed outside of the YMCA. The Co-PI and subject will work together to determine the subject's desired mode and intensity of physical activity, and then construct an exercise prescription to meet current AACE and ACSM physical activity guideline recommendations.

ELIGIBILITY:
Inclusion Criteria

1. Adults age 18 years or older
2. Obese (BMI ≥30 kg/m2), after taking into account age, gender, ethnicity, fluid status, and muscularity
3. Stage of Change Readiness.(Preparation, Action, or Maintenance)
4. Pre-participation Screening based on the ASCM 2015 guidelines
5. Own a functioning Smart phone compatible with CardioCoach VO2 Max app

Exclusion Criteria:

1. Any long-term disease that would interfere with their ability to exercise safely for eg Stroke with extremity weakness
2. Pregnancy
3. Musculoskeletal disorder that prohibits exercise

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-12-05 (Actual); Primary Completion 2020-02-10 (Actual); Study Completion 2020-02-10 (Actual)

PRIMARY OUTCOMES:
Changes in Cardiorespiratory Fitness | 6 Months
  To evaluate whether exercise feedback will effect subjects' Cardiorespiratory Fitness through implementation of a proposed model of Intensive Behavioral Therapy for Obesity utilizing CardioCoachCO2, CardioCoach VO2 Max app, and H10 HR sensors to provide exercise feedback through comparison of VO2Max and VO2Peak to age and sex match norms. Statistical analysis will be performed on VO2Max,VO2Peak, and maximal MET level obtained during a graded exercise test, from baseline and following 6 months of exercise conditioning to determine if a statistically significant or clinically significant change (improvement of 1 MET) which has demonstrated a 12% decrease in all cause morality.

SECONDARY OUTCOMES:
Changes in BMI | 6 Months
  To evaluate whether exercise feedback will effect subjects' changes in BMI consistent with CMS criteria of achieving a weight loss of at least 6.6 lbs (3kg) during the first six months of Intensive Behavioral Therapy for Obesity by comparing BMI from baseline and following 6 months of exercise conditioning through implementation of a proposed model of Intensive Behavioral Therapy for Obesity utilizing CardioCoachCO2, CardioCoach VO2 Max app, and H10 HR sensors to provide exercise feedback.

CONTACTS AND LOCATIONS:
Overall Officials: Debasis Sahoo, MD, Principal Investigator — Attending Physician
Locations (1):
- ClevelandCF South Pointe Hospital, Warrensville Heights, Ohio, United States